CLINICAL TRIAL: NCT07142018
Title: Investigation of the Effect of Hyperbaric Oxygen Therapy on Physical Capacity, Depressive Symptoms, and Quality of Life in Patients With Avascular Necrosis
Brief Title: Investigation of the Effect of Hyperbaric Oxygen Therapy in Patients With Avascular Necrosis
Status: Active, not recruiting | Type: Observational
Sponsor: Dr. Lutfi Kirdar Kartal Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, İsmail Koç, Assistant Prof, Dr. Lutfi Kirdar Kartal Training and Research Hospital
Other Study IDs: Ismail Koc
Record Dates: First submitted 2025-08-19; First posted 2025-08-26 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Avascular Necrosis of Femur Head
MeSH Terms: conditions — Femur Head Necrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Avascular Necrosis: Patients with Avascular Necrosis Undergone Hyperbaric Oxgen

SUMMARY:
Avascular necrosis is a condition that occurs when bone tissue loses sufficient blood flow. This condition causes bone cells to die and, as a result, bone structure to deteriorate.

Hyperbaric oxygen therapy is a treatment method used in patients with avascular necrosis.

Avascular necrosis can significantly affect the quality of life of patients. The aim of this study was to investigate the effects of hyperbaric oxygen therapy on physical capacity, depressive symptoms, and quality of life in patients diagnosed with avascular necrosis.

DETAILED DESCRIPTION:
Avascular necrosis is a condition that occurs when bone tissue loses sufficient blood flow. This condition causes bone cells to die and, as a result, bone structure to deteriorate. It is commonly seen in joints such as the hip, knee, ankle, and shoulder.

Hyperbaric oxygen therapy is a treatment method used in patients with avascular necrosis. In hyperbaric oxygen therapy, patients breathe 100% oxygen under high pressure. This treatment can help treat avascular necrosis by increasing oxygen, promoting new blood vessel formation, reducing inflammation, and facilitating cell repair mechanisms.

Avascular necrosis can significantly affect the quality of life of patients. The effects of avascular necrosis on quality of life can be summarized as follows: Avascular necrosis often causes severe pain and limited mobility in the joint areas. These physical symptoms can prevent patients from performing their daily activities, leading to social isolation and a decline in overall quality of life.

The aim of this study was to investigate the effects of hyperbaric oxygen therapy on physical capacity, depressive symptoms, and quality of life in patients diagnosed with avascular necrosis.

ELIGIBILITY:
Inclusion Criteria:

* Be over 18 years of age,
* Receive hyperbaric treatment,
* Be diagnosed with avascular necrosis,
* Have stage 1-2 avascular necrosis according to the Ficat classification,
* Be able to understand and speak Turkish,
* Be able to read and write,

Exclusion Criteria:

* Having undergone orthopedic surgery on the lower extremities,
* Having cardio-respiratory failure that prevents walking,
* Having a disorder related to the musculoskeletal system other than AVN
* Having a diagnosis of avascular necrosis classified as stage 3-4 according to the Ficat classification
* Presence of varicose veins,
* Presence of urinary stress incontinence,
* Presence of systemic or rheumatological disease,
* Pregnancy,
* Refusal to participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with Avascular Necrosis
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2025-08-19 (Actual); Primary Completion 2025-08-25 (Estimated); Study Completion 2025-08-27 (Estimated)

PRIMARY OUTCOMES:
tinetti performance oriented mobility assessment measure | 1 week
  The Tinetti assessment tool is an easily administered task-oriented test that measures an older adult's gait and balance abilities. Scoring: A three-point ordinal scale, ranging from 0-2. "0" indicates the highest level of impairment and "2" the individuals independence.
Beck Depression Inventory | 1 week
  It is a 21-item, self-report rating inventory that measures characteristic attitudes and symptoms of depression.
Short form 36 | 1 week
  SF-36 is a set of generic, coherent, and easily administered quality-of-life measures. These measures rely upon patient self-reporting and have been widely used.

CONTACTS AND LOCATIONS:
Locations (1):
- Kartal Dr Lutfi Kirdar City Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No